CLINICAL TRIAL: NCT03409575
Title: Efficacy of Two Different Method of Neuromuscular Electrical Stimulation on Quadriceps Strength, Fatigue and Physical Function in Geriatric Population
Brief Title: Efficacy of Neuromuscular Electrical Stimulation in Geriatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sevim ACARÖZ CANDAN (Other)
Collaborators: Scientific Researches Project Coordination Department of Ordu University (Unknown)
Responsible Party: Sponsor-Investigator, Sevim ACARÖZ CANDAN, Head of Department of Physiotherapy and Rehabilitation, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AR-1665
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Age-Related Atrophy; Physical Disorder
Keywords: neuromuscular electrical stimulation; geriatric population; physical function; quadriceps; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 minutes stimulation (Other): The biphasic, symmetrical waveform will be used. The 100 Hz current will be applied for 5 minutes.
  Interventions: Other: 5 minutes stimulation
- 10 minutes stimulation (Other): The biphasic, symmetrical waveform will be used. The 100 Hz current will be applied for 10 minutes.
  Interventions: Other: 10 minutes stimulation

INTERVENTIONS:
Other: 5 minutes stimulation — Before the NMES application, warming exercises will be performed on the lower extremity muscles for 5 minutes. NMES will be administered through Compex device (Physio, Chattanooga Corporation, Chattanooga, U.S.A.). Quadriceps will be stimulated bilaterally for 3 sessions per week for 6 weeks (totally 18 sessions). Four electrodes will be used on the femoral nerve, and motor points of the rectus femoris, vastus medialis, lateralis.The biphasic, symmetrical waveform will be used. The 100 Hz current will be applied for 5 minutes by 5 sec on: 15 sec off and than the muscle will be rested for 10 minutes. 5 minutes of NMES will be made in 4 sets. Fifteen contractions will be received at each set. The intensity of the current will be increased until the visible contraction is taken.
  Arms: 5 minutes stimulation
Other: 10 minutes stimulation — Before the NMES application, warming exercises will be performed on the lower extremity muscles for 5 minutes. NMES will be administered through Compex device (Physio, Chattanooga Corporation, Chattanooga, U.S.A.). Quadriceps will be stimulated bilaterally for 3 sessions per week for 6 weeks (totally 18 sessions). Four electrodes will be used on the femoral nerve, and motor points of the rectus femoris, vastus medialis, lateralis.The biphasic, symmetrical waveform will be used. The 100 Hz current will be applied for 10 minutes by 5 sec on: 15 sec off and than the muscle will be rested for 10 minutes. 10 minutes of NMES will be made in 2 sets. Thirty contractions will be received at each set. The intensity of the current will be increased until the visible contraction is taken.
  Arms: 10 minutes stimulation

SUMMARY:
The decline in physical function and strength was seen by the nature of aging. The older adults often complain of fatigue. For these reasons, proper rehabilitation approaches should be used to ensure healthy life and to keep the quality of life at the highest possible level by minimizing the decline seen with aging process. Exercise programs and Neuromuscular Electrical Stimulation (NMES) are applied in rehabilitation to restore muscular strength and improve physical performance. NMES is used to prevent the atrophy of nonuse, to increase joint range of motion, to re-educate muscle, to regulate spasticity, to replace orthosis, to improve motor involvement of muscle fibers. Despite the use of NMES for strengthening in the clinics, the application parameters and methods should be discussed. The frequency, the pulse duration, the on / off time, the amplitude, the waveform of the current and the application time vary between the studies. For geriatric populations, it is recommended that the highest intensity, biphasic symmetrical currents with a frequency in the range of 50-100 Hz, for 100-400 μs, can be pulsed for ideal amplification. NMES is usually practiced by physiotherapists continuously for 20 minutes in to strengthen. However, in recent studies, it has been shown that continuous application of a single-session 100 Hz current for 20 minutes leads to intense fatigue and after a while the effect of the strengthening of the current has been removed. Therefore, intermittent applications have been proposed instead of continuous applications for 20 minutes. Considering the fragility and the presence of sarcopenia in the geriatric population, NMES applications should be preferred in which rest periods are given instead of continuous application for 20 minutes. In the literature, there is no study showing the effect of NMES on Quadriceps strength, fatigue and physical function by using quadriceps stimulation for 20 minutes using different stimulation periods.Therefore, in this study, will be investigated the possible effects of two different methods of NMES on Quadriceps strength, fatigue and physical function.

ELIGIBILITY:
Inclusion Criteria includes

* age 60 years or older
* be able to climb one floor of stairs independently
* not participate in an exercise program to increase strength or physiotherapy programme.

Exclusion Criteria:

* having a medical condition in which NMES training is contraindicated
* having a cognitive impairment
* having implanted cardiac pacemaker

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Timed up and go test | 2 minutes
  This test will be used to measure the progress of balance, sit to stand, and walking. The participants stands up upon therapist's command walks 3 meters, turns around, walks back to the chair and sits down.
  The time stops when the patient is seated. Time will be recorded.
30-Second Chair Stand Test | 30 second
  The 30CST is a measurement that assesses functional lower extremity strength in older adults. The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand.The score is the total number of stands within 30 seconds (more than halfway up at the end of 30 seconds counts as a full stand). Incorrectly executed stands are not counted.
6 minute walk test | 6 minute
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The participant walk for 6 minutes on 30 meter long way. The total distance will be recorded at the end of the test.

SECONDARY OUTCOMES:
Grip Strength | 5 minutes
  The patient wiil squeeze the dynamometer as the arm is adjacent to the body, the elbow is at 90 ° flexion, the forearm is in the neutral position and the wrist is at 0-30 ° extension. After the test is repeated three times, the highest score will be recorded. The test will only be done for the dominant hand.
Berg Balance Scale | 10 minutes
  The balance will be evaluated observational during 14 different balance activities. A five-point scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. It's minimum and maximum scores ranged between 0 and 56.
  Interpretation: 41-56 = low fall risk 21-40 = medium fall risk 0 -20 = high fall risk
Strength of Quadriceps muscle | 5 minutes.
  Lafayette manuel muscle tester will be used to determine the strength of the Quadriceps. The strength will be evaluated bilaterally three times and then the maximum value will be recorded.
Short Physical Performance Battery | 3 minutes
  The battery is an objective assessment tool for evaluating lower extremity functioning in older persons. The battery is scored between 0-12 scores according to the balance, chair stand test performance and gait speed of the participant.
Fatigue Severity Scale | 5 minutes
  The 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Each item is scored between1 and 7. A low value (e.g., 1) indicates strong disagreement with the statement, whereas a high value (e.g., 7) indicates strong agreement. A total score of 36 or more suggests that you may be suffering from the fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim A CANDAN, Principal Investigator — Ordu University
Locations (2):
- Turkey (Türkiye) (2):
  - Sevim ACARÖZ CANDAN, Ordu, Altinordu
  - Sevim ACARÖZ CANDAN, Ordu

IPD SHARING:
Plan to Share IPD: No